CLINICAL TRIAL: NCT01162005
Title: Therapeutic Effect of Tacrolimus on Primary Nephrotic Syndrome in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Il Soo Ha, Study chair, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INS-Tacrobell; INS-Tacrobell-Pediatrics (Other: Seoul National University Hospital)
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Results first posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2018-09

CONDITIONS: Nephrotic Syndrome
Keywords: Primary Nephrotic syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus (Experimental): Tacrobell
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — dosage : 0.1-0.2 mg/kg/day divided two target trough level : 5 - 10 ng/mL Total duration (tacrolimus) : 1 year
  Other Names: Trcrobell

SUMMARY:
To determine the efficacy of tacrolimus in the management of NS(nephrotic syndrome) , the investigators designed this prospective study. The investigators will enroll 100 children with NS(frequent relapse steroid dependent NS, steroid resistance NS) who will be treated with tacrolimus (0.1-0.2 mg/kg/day in two divided doses over 12 h adjusted to a trough level between 5 and 10 ng/ml) for 12 months in combination with low-dose steroids. Other therapies will be included angiotensin-converting enzyme inhibitors, antihypertensive drugs, multivitamins and lipid-lowering agents.

Follow-up is every second week for the first 4 weeks, then monthly. After initiation of tacrolimus therapy, blood was drawn each visit to determine tacrolimus trough levels.

DETAILED DESCRIPTION:
Subsequently , monthly measurements were made until stable levels of tacrolimus were achieved. Urine was analyzed for proteinuria at each visit. Serum creatinine, glucose, albumin and alanine aminotransferase were measured and complete blood counts were obtained at each visit during the study.

ELIGIBILITY:
Inclusion Criteria:

* Frequent relapse nephrotic syndrome
* steroid resistance nephrotic syndrome

Exclusion Criteria:

* secondary nephrotic syndrome
* estimated glomerular filtration rate < 60 mL/min/1.73m2
* with active hepatitis

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2010-07; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ILSOO Ha, MD, PhD, Study Chair — Seoul National Children's Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 2010 to August 2013, children with refractory NS were enrolled.
  It was conducted at three centers in Korea after obtainment of informed consent.
  ( Seoul National University Children's Hospital, Samsung Medical Center, Asan Medical Center Children's Hospital)
Groups:
- SDNS/FRNS Group: Indicative of two or more relapses during tapering or within 14 days of stopping steroid therapy or more than four relapses within one year or at least two within six months
  SDNS: steroid-dependent nephrotic syndrome; FRNS: frequent-relapsing nephrotic syndrome;
- SRNS Group: Absence of remission after four weeks of steroid therapy SRNS: steroid-resistant nephrotic syndrome
Period: Overall Study
Arm/Group | SDNS/FRNS Group | SRNS Group
Started | 44 | 33
Completed | 44 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SDNS/FRNS Group: SDNS: steroid dependent nephrotic syndrome FRNS: frequent relapsing nephrotic syndrome
  Indicative of two or more relapses during tapering or within 14 days of stopping steroid therapy or more than four relapses within one year or at least two within six months
- SRNS Group: SRNS: steroid resistant nephrotic syndrome
  Absence of remission after four weeks of steroid therapy.
- Total: Total of all reporting groups
Arm/Group | SDNS/FRNS Group | SRNS Group | Total
Number analyzed (Participants) | 44 | 33 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (4.2) | 7.9 (4.2) | 9.9 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 35 | 19 | 54

OUTCOME MEASURES:

1. Primary Outcome: Remission Rate
Description: Complete remission at 12 months Per KDIGO clinical practice guideline for glomerulonephritis (2012): Complete remission (CR), urine protein creatinine ratio below 200mg/g (20mg/mmol) or 1+ of protein on urine dipstick for 3 consecutative days
Time Frame: 12-month treatment period
Measure: Count of Participants; unit: Participants
Groups:
- SDNS/FRNS: Indicative of two or more relapses during tapering or within 14 days of stopping steroid therapy or more than four relapses within one year or at least two within six months
- SRNS: Absence of remission after four weeks of steroid therapy
Arm/Group | SDNS/FRNS | SRNS
Number analyzed (Participants) | 44 | 33
Participants | 34 | 13
Statistical Analysis 1: Comparison: SDNS/FRNS vs SRNS; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

2. Secondary Outcome: Duration of Remission
Description: Mean duration of remission
Time Frame: 12-month treatment period
Measure: Mean (Standard Deviation); unit: months
Groups:
- SDNS/FRNS Group: Indicative of two or more relapses during tapering or within 14 days of stopping steroid therapy or more than four relapses within one year or at least two within six months
- SRNS Group: Absence of remission after four weeks of steroid therapy
Arm/Group | SDNS/FRNS Group | SRNS Group
Number analyzed (Participants) | 44 | 33
months | 4.6 (2.9) | 4.0 (3.2)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | SDNS/FRNS Group | SRNS Group
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/44 | 4/33
Other Adverse Events (participants affected / at risk) | 3/44 | 16/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SDNS/FRNS Group (N=44) | SRNS Group (N=33)
Decreased renal function (Renal and urinary disorders) | 0 (0) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SDNS/FRNS Group (N=44) | SRNS Group (N=33)
Transient glycosuria (Blood and lymphatic system disorders) | 3 (3) | 8 (8)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Gastrointestinal trouble (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 2 (2)
Transient hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Itching sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes